CLINICAL TRIAL: NCT06657157
Title: Peripheral Neuropathy in Patients Receiving Pembrolizumab and Enfortumab Vedotin as First Line Treatment for Metastatic or Locally Advanced Urothelial Carcinoma. An Investigator-Initiated, Prospective, Multicenter, Non-Interventional Trial.
Brief Title: Peripheral Neuropathy in Patients Receiving Enfortumab Vedotin and Pembrolizumab as First Line Treatment for Metastatic or Locally Advanced Urothelial Carcinoma
Acronym: P-EVOLUTION
Status: Recruiting | Type: Observational
Sponsor: Comprehensive Cancer Center Munich (CCCM) (Other)
Collaborators: Department of Urology, LMU University Hospital Munich, Munich, Germany (Unknown); Department of Urology, TUM Klinikum rechts der Isar, Munich, Germany (Unknown)
Responsible Party: Principal Investigator, Can Aydogdu, MD, Principal Investigator, Comprehensive Cancer Center Munich (CCCM)
Other Study IDs: P-EVOLUTION
Record Dates: First submitted 2024-10-19; First posted 2024-10-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Urothelial Cancer
Keywords: enfortumab vedotin; Pembrolizumab; peripheral neuropathy; metastatic urothelial carcinoma; advanced urothelial carcinoma
MeSH Terms: conditions — Peripheral Nervous System Diseases; Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The P-EVOLUTION trial is a prospective, multicenter, non-interventional observational study aimed at investigating peripheral neuropathy in patients receiving first-line treatment for metastatic or locally advanced urothelial carcinoma with enfortumab vedotin (EV) and pembrolizumab (P). Conducted at two German university hospitals, the study will track the incidence and severity of peripheral neuropathy, its impact on quality of life, and treatment regimen adjustments due to side effects. Approximately 80 patients are expected to be enrolled over one year.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, ≥18 years of age at the time of signing the informed consent form (ICF)
* Patients with histologically confirmed metastatic or locally advanced, unresectable urothelial carcinoma
* Patients who did not receive any systemic treatment for their laUC or mUC (treatment-naïve)
* Patients who are able to receive enfortumab vedotin and pembrolizumab according to the respective medicinal product information

Exclusion Criteria:

* Patients with contraindications for enfortumab vedotin and/or pembrolizumab
* Patients who have received a systemic therapy for their laUC or mUC (e.g. platinum-based chemotherapy, checkpoint-inhibitors)
* Patients who have previously been treated with enfortumab vedotin, other MMAE-based antibody-drug-conjugates or PD-(L)1-checkpoint inhibitors
* Patients who received neoadjuvant or adjuvant platinum-based chemotherapy <12 months ago

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting the eligibility criteria and are treated at the tertiary care centers LMU Munich and TUM Munich.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of peripheral neuropathy ≥ CTCAE grade 2 | baseline, week 18, week 36, week 52, and End of Treatment (defined as the administration of the last dose of EV/P)
  Incidence of peripheral neuropathy ≥ grade 2 at baseline, week 18, week 36, week 52, and at End of Treatment (defined as the administration of the last dose of EV/P) assessed by the Patient Neurotoxicity Questionnaire (PNQ)

SECONDARY OUTCOMES:
Change of degree of sensory, motor and/or autonomic peripheral neuropathy applying the EORTC-CIPN20 questionnaire | Baseline, week 18, week 36, week 52, and End of Treatment (defined as the administration of the last dose of EV/P)
  A higher EORTC-CIPN20 score indicates a worse degree of neuropathy.
Change of Quality of life (QoL) applying the FACT/GOG-NTX questionnaire | Baseline, week 18, week 36, week 52, and End of Treatment (defined as the administration of the last dose of EV/P)
  An higher FACT/GOG-NTX score indicates a better QoL.
Change of neuropathic pain applying the Neuropathic Pain Symptom Inventory (NPSI) questionnaire | Baseline, week 18, week 36, week 52, and End of Treatment (defined as the administration of the last dose of EV/P)
  A higher NPSI score indicates more neuropathic pain.
Change of depression based on the Allgemeine Depressionsskala (ADS) | Baseline, week 18, week 36, week 52, and End of Treatment (defined as the administration of the last dose of EV/P)
  A higher ADS value indicates higher degree of depression.
Time to onset of peripheral neuropathy ≥ CTCAE grade 2 | From the administration of the first dose of EV/P to the end of treatment (defined as the administration of the final dose of EV/P), which is expected to occur after approximately one year.
Number of dose reductions, delays or treatment discontinuation due to peripheral neuropathy or other adverse events | From the administration of the first dose of EV/P to the end of treatment (defined as the administration of the final dose of EV/P), which is expected to occur after approximately one year.
Number of cycles of EV + P administered | From the administration of the first dose of EV/P to the end of treatment (defined as the administration of the final dose of EV/P), which is expected to occur after approximately one year.
Change in nerve conduction studies, as measured by neurography, in the right tibial (motor) nerve | Baseline, Week 18, End of Treatment (defined as the administration of the final dose of EV/P)
  A higher nerve conduction velocity indicates a faster transmission of electrical signal along the nerve. And vice versa.
Change in nerve conduction studies, as measured by neurography, in the right sural (sensory) nerve | Baseline, Week 18, End of Treatment (defined as the administration of the final dose of EV/P)
  A higher nerve conduction velocity indicates a faster transmission of electrical signal along the nerve. And vice versa.
Changes in hand force as measured with a Martin-Vigorimeter | Baseline, Week 18, End of Treatment (defined as the administration of the final dose of EV/P)
Changes in sensory perception using a monofilament test | Baseline, Week 18, End of Treatment (defined as the administration of the final dose of EV/P)
Overall survival | From administration of first dose to date of death of any cause, assessed for up to 60 months
  defined as the time from administration of the first dose to date of death due to any cause
real world Progression free survival (rw-PFS) | From administration of the first dose of EV/P to the first documented disease progression, as determined by the investigator, or to death from any cause, whichever occurs first, assessed up to 60 months.
  rw-PFS, defined as the time from the administration of the first dose of EV/P to the first documented disease progression, as determined by the investigator, or to death from any cause, whichever occurs first, assessed up to 60 months.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Urology, LMU University Hospital, Ludwig-Maximilians-University Munich, Munich, Bavaria
  - Department of Urology, Klinikum rechts der Isar, Technical University Munich, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided